CLINICAL TRIAL: NCT04044131
Title: A Phase 2, Randomized, Placebo Controlled Study to Evaluate the Efficacy, Tolerability and Safety of Metabolic Cofactor Supplementation in Alzheimer's Disease (AD) And Parkinson's Disease (PD) Patients
Brief Title: Metabolic Cofactor Supplementation in Alzheimer's Disease (AD) and Parkinson's Disease (PD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: ScandiBio Therapeutics AB (Industry); Alanya Alaaddin Keykubat University (Other); Sahlgrenska University Hospital (Other); KTH Royal Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Lutfu Hanoglu, MD, Professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Metabolic Cofactor Study
Record Dates: First submitted 2019-07-17; First posted 2019-08-05 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Alzheimer Disease; Parkinson Disease
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease | interventions — Sorbitol

STUDY DESIGN:
Intervention Model Description: A total of 60 Alzheimer's and 60 Parkinson's disease patients will be randomized on a 2:1 basis to the cofactor mixture or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Subjects in active treatment will receive dietary supplementation with N-acetylcysteine, L-carnitine tartrate, nicotinamide riboside, and serine, administered as a mixture.
  Interventions: Drug: Metabolic Cofactor Supplementation
- Placebo Arm (Placebo Comparator): Subjects will take a mixture of placebo as powder dissolved in water by mouth.
  Interventions: Drug: Sorbitol

INTERVENTIONS:
Drug: Metabolic Cofactor Supplementation — Dietary supplement consisting of serine, L-carnitine tartrate, N-acetylcysteine and nicotinamide riboside. Subjects in active treatment will receive dietary supplementation with N-acetylcysteine, L-carnitine tartrate, nicotinamide riboside, and serine, administered as a mixture. Half dosage of the co-factors will be given for two weeks (one dose taken just after dinner), and full dosage for 8 weeks (two equal doses taken just after breakfast and dinner).
  Arms: Treatment Arm
Drug: Sorbitol — As placebo, sorbitol (5g) flavoured with strawberry aroma and colouring agent will be given.
  Arms: Placebo Arm

SUMMARY:
This double-blind, randomized, placebo-controlled, investigator-initiated, multi-centre trial aims to establish metabolic improvements in AD and PD subjects by dietary supplementation with cofactors N-acetylcysteine, L-carnitine tartrate, nicotinamide riboside and serine. Concomitant use of pivotal metabolic cofactors via simultaneous dietary supplementation will stimulate to enhance hepatic β-oxidation and this study's hypothesis is that this will result in increased mitochondrial activity in human brain cell-types.

DETAILED DESCRIPTION:
In this study, investigators aim to activate mitochondria of brain cell-types in AD and PD patients by increasing the hepatic, plasma and brain levels of pivotal metabolic cofactors via simultaneous dietary supplementation of serine, L-carnitine, N-acetylcysteine (NAC) and nicotinamide riboside (NR).

The study is based on a three-step strategy to activate the mitochondria in human brain cells: (1) The investigators will use L-carnitine tartrate to enhance the transport of fatty acids across the mitochondrial membrane (by forming a long chain acetylcarnitine ester and being transported by carnitine palmitoyltransferase [CPT] I and CPT II) and to stabilize acetyl-CoA and coenzyme A levels. (2) Nicotinamide riboside, precursor of NAD+ will be included to boost the level of hepatic β-oxidation of fatty acids in mitochondria. Decreased electron transport chain function combined with impaired rates of fatty acid β-oxidation leads to the accumulation of incomplete products of β-oxidation, which combined with increased levels of reactive oxygen species (ROS), contribute to insulin resistance. Nicotinamide riboside stimulates the transfer of fatty acids from cytosol to mitochondria, similar to L-carnitine tartrate. (3) Two glutathione precursors, serine and N-acetylcysteine, will be included to increase glutathione levels in the hepatocytes. Increased glutathione levels will also protect against free radical-mediated oxidative stress generated by the increased β-oxidation of fatty acids in mitochondria.

Previous studies showed that each agent is able to activate mitochondria separately and a proof-of-concept study using serine supplementation, and a phase I study using this three-step approach resulted in a significant decrease in plasma metabolites associated with mitochondrial dysfunction without significant side effect. The novel design with this study is to give the L-carnitine, NR, serine and NAC as a cocktail. Based on investigators' earlier results, that this will improve the efficacy of the intervention.

The study population will consist of 60 Alzheimer's and 60 Parkinson's disease patients. Eligible subjects must have signed an informed consent, meet all inclusion criteria and have none of the exclusion criteria listed below. Patients will be randomized on a 2:1 basis to the cofactor mixture or placebo in two different centres.

The subjects will take a mixture of cofactors or matching placebo as powder dissolved in water by mouth. Subjects in active treatment will receive dietary supplementation with N-acetylcysteine, L-carnitine tartrate, nicotinamide riboside, and serine, administered as a mixture. Half dosage of the co-factors will be given for two weeks (one dose taken just after dinner), and full dosage for 8 weeks (two equal doses taken just after breakfast and dinner). Patients who cannot tolerate taking full dose may continue the study with half dose (i.e. one dose taken just after dinner). Patients who cannot tolerate the study agents will be withdrawn from the study.

Active treatment duration will be 12 weeks for each subject and the total study duration is estimated as 6 months. Study comprises four clinical visits; (1) a screening visit, (2) randomization visit, (3) treatment visit and (4) end of treatment visit. At visit 1 and visit 4, all procedures including clinical and physical examination, adverse events recording, MRI volumetric and rest-state fMRI, determination of the motor, cognitive and behavioral functions using clinical scales, biochemical, omic and oral/gut microbiota analysis will be done. At visit 2, eligible study subjects will be randomized to active therapy or placebo groups and study agents will be dispensed. At visit 3, clinical and physical examination, determination of the motor, cognitive and behavioural functions using clinical scales, laboratory safety parameters, omic and oral/gut microbiota analysis will be repeated as in Visit 1. After the visit 4, participants will stop taking study agents.

A subject will be considered as having completed the study if he/she has completed all assessments at the End of Treatment Visit (Visit 4) and has been followed up until 12 weeks after initiation of the study drugs.

Statistics for the primary outcome parameter will be analysed by Mann-Whitney U test or t-test depending on the results of the normality test. For the secondary outcome parameters, one-way repeated measures ANOVA will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with Parkinson's Disease (Hoehn Yahr 2-4, age >18 years) or men and women diagnosed with Alzheimer's Disease. Include patients older than 50 years with mild to moderate Alzheimer's disease according to ADAS-cog (Alzheimer's Disease Assessment Scale-cognitive subscale; ADAS≥12) and the Clinical Dementia Rating Scale Sum of Boxes (CDR-SOB; CDR≤2).
* Patients with stable treatments and clinical course

Exclusion Criteria:

* Inability or unwillingness to give written informed consent
* History of stroke, severe brain trauma, toxic drug exposure
* Neurological examination which indicate to Parkinson-Plus syndrome (i.e., pyramidal, cerebellar and autonomic dysfunction findings and gaze paralysis) for PD
* Uncontrolled Type 1 or type 2 diabetes
* Diarrhea (defined as more than 2 stool per day) within 7 days before enrolment
* Chronic kidney disease with an estimated glomerular filtration rate <60 ml/min/1.73m2
* Significant cardiovascular co-morbidity (i.e. heart failure, documented coronary artery disease, valvular heart disease)
* Patients with active bronchial asthma
* Patients with phenylketonuria (contraindicated for NAC)
* Patients with histamine intolerance
* Clinically significant TSH level outside the normal range (0.04-6 mU/L)
* Known allergy for substances used in the study
* Concomitant medication use: Self-administration of dietary supplements such as any vitamins, omega-3 products, or plant stanol/sterol products within 1 month; Use of an antimicrobial agent in the 4 weeks preceding randomization
* Active smokers consuming >10 cigarettes/day
* Alcohol consumption over 192 grams for men and 128 grams for women per week
* Patients considered as inappropriate for this study for any reason (patients unable to undergo MRI study, noncompliance etc.)
* Active participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Mini Mental State Examination (MMSE) | 4 weeks and 12 weeks
  The change in Mini Mental State Examination (MMSE) scores between the placebo and the treatment arms in AD patient from baseline to 4 weeks and 12 weeks. MMSE is global cognitive evaluation scale for AD patients. It consists of eleven questions and is evaluated over 30 points. It is normal between 24-30 points.
Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog) | 4 weeks and 12 weeks
  The change in Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog) scores between the placebo and the treatment arms in AD patients from baseline to 4 weeks and 12 weeks. ADAS-cog is cognitive evaluation scale for AD patients. ADAS-Cog includes 11 tasks that include both subject-completed tests and observer-based assessments. Together these tasks assess the cognitive domains of memory, language, and praxis. The ADAS-cog is scored between 0-70 and high scores indicate poor status.
Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) | 4 weeks and 12 weeks
  The change in Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) scores between the placebo and the treatment arms in AD patients from baseline to 4 weeks and 12 weeks. ADCS-ADL is daily life activity evaluation scale for AD patients. This is a questionnaire structured to evaluate functional capacity in AD patients. It is scored between 0-78 and low scores indicate addiction. It is applied to the patient's relatives.
Unified Parkinson's Disease Rating Scale (UPDRS) | 4 weeks and 12 weeks
  The change in Unified Parkinson's Disease Rating Scale (UPDRS) scores between the placebo and the treatment arms in PD patients from baseline to 4 weeks and 12 weeks. UPDRS is motor evaluation scale for PD patients. The UPDRS is used to follow the longitudinal course of Parkinson's disease. UPDRS has four parts: Part I (non-motor experiences of daily living), Part II (motor experiences of daily living, Part III (motor examination) and Part IV (motor complications). The first part 4, the second part 13, the third part 14 and the fourth part consists of 11 items. Each item scored between 0 (none) and 4 (heaviest). A score of 147 on the UPDRS scale represents the worst (total disability) with a score of zero representing (no disability).

SECONDARY OUTCOMES:
Volumetric Magnetic resonance Imaging (MRI) and resting state functional magnetic resonance imaging (rest-fMRI) | 12 weeks
  The change in central nervous system atrophy and resting state network activity between the placebo and the treatment arms in AD and PD patients from baseline to 12 weeks.
Neuropsychiatric Inventory (NPI) | 4 weeks and 12 weeks
  The change in Neuropsychiatric Inventory (NPI) scores between the placebo and the treatment arms in AD and PD patients from baseline to 4 weeks and 12 weeks. NPI is behavioural evaluation scale for PD and AD patients. It is evaluated delusions, hallucinations, agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, irritability/lability, aberrant motor activity, night-time behavioral disturbances and appetite, eating abnormalities. It is applied to the patient's relatives. If the patient's relative verifies the presence of that symptom, it is continued with more specific questions of that area. Subsequently, multiplying the numerical values given for the frequency (1 rare-4 very frequent) and severity (1 mild-3 severe) of the symptom constitutes the score of that item. The maximum score can be 144. For each item, the distress caused by that symptom for the relative of the patient is also calculated over 6 points (0 none-5 very severe).
Montreal Cognitive Assessment (MoCA) | 4 weeks and 12 weeks
  The change in Montreal Cognitive Assessment (MoCA) scores between the placebo and the treatment arms in PD patients from baseline to 4 weeks and 12 weeks. MoCA is global cognitive evaluation scale for PD patients. The MoCA evaluates different types of cognitive abilities. These include orientation, short-term memory/delayed recall, executive function/visuospatial ability, language abilities, abstraction, animal naming, attention, clock-drawing test. Scores on the MoCA range from zero to 30, with a score of 26 and higher generally considered normal.
Changes in serum omic profile from baseline | 4 weeks and 12 weeks
  The change in omic profile between the placebo and the treatment arms in PD an AD patients from baseline to 4 weeks and 12 weeks. Neurodegenerative diseases are affected by a combination of genetic, epigenetic and environmental factors. Omic studies are useful for deciphering the molecular landscape of neurodegenerative diseases. Omic data collected from both the PD and AD patient group will be used to identify molecular networks, biomarkers, and possible therapeutic targets through system biology. The aim of this study is to determine possible subtypes of disease based on the patients' response to treatment and to translate the network-based findings into clinically applicable tools for personalized medical practice. Serum omic analysis will include generation of untargeted omics data in Sweden. Biomarkers will be analysed by proximity extension and proximity ligation technologies (PEA and PLA) providing assays with high specificity and sensitivity in complex biological matrices.
Microbiota analysis | 4 weeks and 12 weeks
  The change in gut microbiota between the placebo and the treatment arms in PD an AD patients from baseline to 4 weeks and 12 weeks. Faeces and saliva samples will be collected to assess changes in gut microbiota. Instructions on specimen collection will be given during the first visit. Microbiota will be assessed using shot-gun metagenomic techniques.
Monitoring of adverse events | 1 week, 4 weeks and 12 weeks
  This process aiming to monitoring of adverse events of metabolic cofactor supplementation. Adverse events and serious adverse events will be monitored continuously and all adverse events that occur at any time during the study will be reported in Case Report Forms. Any symptoms of intestinal discomfort or other side effects will be carefully recorded and all study subjects will be informed to contact (by phone or text message) the investigators immediately if they experience any symptoms of discomfort or any side effects during the intervention period.
Change in heart rate from baseline | 1 week, 4 weeks and 12 weeks
  Heart rate will be measured at every visit to evaluate safety of metabolic cofactor supplementation.
Change in blood pressure from baseline | 1 week, 4 weeks and 12 weeks
  Blood pressure will be measured at every visit to evaluate safety of metabolic cofactor supplementation.
Change in waist and hip circumference from baseline | 1 week, 4 weeks and 12 weeks
  Waist and hip circumference will be measured at every visit to evaluate safety of metabolic cofactor supplementation.
Change in body weight from baseline | 1 week, 4 weeks and 12 weeks
  Body weight will be measured at every visit to evaluate safety of metabolic cofactor supplementation.
Change of complete blood count from baseline | 4 weeks and 12 weeks
  Complete blood count includes number of blood cells and concentration of hemoglobin. Complete blood count will be performed to measure possible toxic effects of the metabolic cofactor supplementation on hematological system.
Changes in liver function tests (alkaline phosphatase (ALP), alanine aminotransferase (ALT), Aspartate aminotransferase (AST), gamma-glutamyl transferase (GGT), total and direct Bilirubin, Albumin) from baseline | 4 weeks and 12 weeks
  Liver function tests (AST, ALT, GGT, total and direct Bilirubin, Albumin) will be performed to measure possible toxic effects of the metabolic cofactor supplementation on liver function.
Changes in blood lipid levels (total cholesterol (TC), triglyceride (TG), low density lipoprotein (LDL-C), high density lipoprotein (HDL-C)) from baseline | 4 weeks and 12 weeks
  Blood lipid levels (total cholesterol (TC), triglyceride (TG), low density lipoprotein (LDL-C), high density lipoprotein (HDL-C)) will be evaluated to measure possible toxic effects of the metabolic cofactor supplementation.
Changes in kidney function tests (creatinine, urea, urate, sodium, potassium) from baseline | 4 weeks and 12 weeks
  Kidney function tests (creatinine, urea, urate, sodium, potassium) will be performed to measure possible toxic effects of the metabolic cofactor supplementation on kidney function.
Changes in creatinine kinase (CK) level from baseline | 4 weeks and 12 weeks
  Creatinine kinase (CK) level will be evaluated to measure possible toxic effects of the metabolic cofactor supplementation.
Change in thyroid-stimulating hormone (TSH) level from baseline | 4 weeks and 12 weeks
  Thyroid-stimulating hormone (TSH) level will be evaluated to measure possible toxic effects of the metabolic cofactor supplementation.
Change in blood insulin level from baseline | 4 weeks and 12 weeks
  Blood insulin level will be evaluated to measure possible toxic effects of the metabolic cofactor supplementation.
Change in glycated haemoglobin (HbA1c) level from baseline | 4 weeks and 12 weeks
  HbA1c level will be evaluated to measure possible toxic effects of the metabolic cofactor supplementation.
Changes in blood glucose levels from baseline | 4 weeks and 12 weeks
  Blood glucose levels will be evaluated to measure possible toxic effects of the metabolic cofactor supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Lutfu Hanoglu, MD, PhD, Principal Investigator — Medipol University; Burak Yulug, MD, PhD, Principal Investigator — Alanya Alaaddin Keykubat University
Locations (2):
- Turkey (Türkiye) (2):
  - Alanya Alaaddin Keykubat University Hospital, Antalya
  - Medipol University Hospital, Istanbul

REFERENCES:
- [Derived] Yulug B, Altay O, Li X, Hanoglu L, Cankaya S, Velioglu HA, Lam S, Yang H, Coskun E, Idil E, Bayraktaroglu Z, Nogaylar R, Ozsimsek A, Yildirim S, Bolat I, Kiliclioglu M, Bayram C, Yuksel N, Tozlu OO, Arif M, Shoaie S, Hacimuftuoglu A, Zhang C, Nielsen J, Turkez H, Boren J, Uhlen M, Mardinoglu A. Multi-omics characterization of improved cognitive functions in Parkinson's disease patients after the combined metabolic activator treatment: a randomized, double-blinded, placebo-controlled phase II trial. Brain Commun. 2025 Jan 6;7(1):fcae478. doi: 10.1093/braincomms/fcae478. eCollection 2025. PMID 39816194
- [Derived] Yulug B, Altay O, Li X, Hanoglu L, Cankaya S, Lam S, Velioglu HA, Yang H, Coskun E, Idil E, Nogaylar R, Ozsimsek A, Bayram C, Bolat I, Oner S, Tozlu OO, Arslan ME, Hacimuftuoglu A, Yildirim S, Arif M, Shoaie S, Zhang C, Nielsen J, Turkez H, Boren J, Uhlen M, Mardinoglu A. Combined metabolic activators improve cognitive functions in Alzheimer's disease patients: a randomised, double-blinded, placebo-controlled phase-II trial. Transl Neurodegener. 2023 Jan 26;12(1):4. doi: 10.1186/s40035-023-00336-2. PMID 36703196